CLINICAL TRIAL: NCT06935422
Title: Role of Cerebroplacental Ratio Discordance at 16-20 Weeks in Predicting Monochorionic Twin Pregnancies' Specific Complications : a Prospective Cohort Study
Brief Title: Role of Cerebroplacental Ratio Discordance at 16-20 Weeks in Predicting Monochorionic Twin Pregnancies' Specific Complications
Acronym: CPR
Status: Recruiting | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Ali Hassan Ali, Director, Ain Shams Maternity Hospital
Other Study IDs: Monochorionic twins
Record Dates: First submitted 2025-03-12; First posted 2025-04-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Monochorionic Twins; Cerebroplacental Ratio
Keywords: Monochorionic twins
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Ultrasound — Measuring cerebroplacental ratio discordance in monochorionic twins at 16-20 Weeks of gestation

SUMMARY:
The purpose of this study is to evaluate the predictive value of CPR discordance at 16-20 weeks in MCDA twin pregnancies in predicting monochorionic-specific complications such as TTTS, TAPS, sFGR and IUFD of one or both fetuses

DETAILED DESCRIPTION:
Monochorionic (MC) twin pregnancies are at a higher risk of perinatal morbidity and mortality because of the risk of developing unique complications. These include twin to twin transfusion syndrome (TTTS), selective fetal growth restriction (sFGR) , twin anemia polycythemia sequence (TAPS) and intrauterine fetal death (IUFD) of one or both fetuses. Therefore, early identification of these conditions is warranted to plan proper perinatal surveillance and management to improve outcome.

Sparse studies have found that inter-twin differences in Doppler ultrasound may occur prior to meeting diagnostic criteria for TTTS, TAPS, sFGR or adverse perinatal outcomes.

This study will try to reveal the potential clinical predictive value of inter-twin cerebroplacental ratio (CPR) discordance in the surveillance of MC twin pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more and able to consent.
* Monochorionic Diamniotic twin pregnancy.
* Discordant inter-twin cerebroplacental ratio at 16-20 weeks of gestation.

Exclusion Criteria:

* Fetal structural malformations or chromosomal abnormalities in any of the twins as detected by anomaly scan antenatally or neonatal examination postnatally (chromosomal abnormalities and some congenital malformations can interfere with normal fetal growth).
* Identified infectious etiologies detected during immediate postnatal examination or during pregnancy (fetal infections can cause FGR ,usually symmetric type particularly if they occur in early gestation).
* Referral after development of Twin to twin transfusion syndrome, twin anemia polycythemia sequence or selective fetal growth restriction.
* Single fetal demise at the time enrollment in the study.
* Conjoint twins.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Monochorionic diamniotic twin pregnancies with discordant cerebroplacental ratio at 16-20 weeks of gestation presenting to Ain Shams University Maternity Hospital for antenatal care.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Development of monochorionic specific complications | From 16-20 weeks of gestation till delivery.
  Monochorionic specific complications include twin to twin transfusion syndrome, twin anemia polycythemia sequence and selective fetal growth restriction

SECONDARY OUTCOMES:
Occurrence of intrauterine fetal death or perinatal mortality of one or both fetuses | From 16-20 weeks of gestation till 7th day of life
  Gestational age upon occurrence of IUFD with clarifying if complications occur in the surviving twin in case of single fetal demise. Time and reason of perinatal mortality for any of the fetuses Wil be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Abdelbaset Abd elkawy, Assistant professor, Study Chair — Ain Shams Maternity Hospital; Haitham Mohsen Elsabaa, Professor, Study Chair — Ain Shams Maternity Hospital; Amr Fathy Abd elkareem, Professor, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Name and email address
Supporting Information: Study Protocol
Time Frame: From 2025 till 2028
Access Criteria: Any researcher, physician or university lecturer Access for full study content

REFERENCES:
- [Background] Jain A, Acharya V, Shettikeri A, Sahana R, Radhakrishnan P. Intertwin discordance in MCA-PI and CPR in the prediction of TTTS progression. 19th world congress in fetal medicine. Ultrasound Obstet Gynecol. 2022;1(1):5-9.
- [Background] Conde-Agudelo A, Villar J, Kennedy SH, Papageorghiou AT. Predictive accuracy of cerebroplacental ratio for adverse perinatal and neurodevelopmental outcomes in suspected fetal growth restriction: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Oct;52(4):430-441. doi: 10.1002/uog.19117. Epub 2018 Sep 5. PMID 29920817
- [Background] Albu AR, Anca AF, Horhoianu VV, Horhoianu IA. Predictive factors for intrauterine growth restriction. J Med Life. 2014 Jun 15;7(2):165-71. Epub 2014 Jun 25. PMID 25408721